CLINICAL TRIAL: NCT06906315
Title: Therapeutic Management of Dexamethasone in Patients Undergoing Endodontics: Randomized Clinical Trial
Brief Title: Dexamethasone Treatment for Patients Undergoing Endodontics
Acronym: (DTPE-RCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Heilyn Nils, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1320-4208; 2025_01/345 (Registry Identifier: Bioethics Committee of Alfonso X el Sabio University, Madrid, Spain)
Record Dates: First submitted 2025-03-16; First posted 2025-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Endodontic Treatment; Pulp Necrosis; Periapical Lesions; Postoperative Pain
Keywords: Endodontic Pain Management; Dexamethasone; Postoperative Pain; Corticosteroids in Endodontics; Visual Analog Scale (VAS)
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment interventional model, where participants were randomly assigned to one of two groups:
  Dexamethasone Group: Received a single 4 mg oral dose of dexamethasone 1 hour before endodontic treatment.
  Ibuprofen Group: Received no preoperative medication but took 400 mg of ibuprofen every 4 hours postoperatively for pain management.
  Both groups underwent the same standardized endodontic procedure, ensuring that the only variable was the pain management intervention.
  This was a single-blind study where participants were blinded to treatment allocation. Randomization was performed in a 1:1 ratio using simple randomization.
  The primary outcome was postoperative pain intensity, measured using the VAS scale at 4, 6, 8, 12, and 24 hours. Secondary outcomes included rescue analgesia use and adverse effects.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Group (Experimental): Participants in this group received a single 4 mg oral dose of dexamethasone 1 hour before undergoing endodontic treatment. No additional preoperative analgesics were administered. Standard endodontic procedures, including local anesthesia, were performed. Post-treatment, no routine analgesic medication was provided unless additional pain relief was required. Pain intensity was assessed at 4, 6, 8, 12, and 24 hours using the Visual Analog Scale (VAS) to evaluate the efficacy of preoperative dexamethasone in controlling postoperative pain and inflammation.
  Arm 2
  Interventions: Drug: Dexamethasone 4 mg
- Ibuprofen Group (Active Comparator): Participants in this group received no preoperative medication but were prescribed 400 mg of ibuprofen every 4 hours postoperatively for pain management. The same standard endodontic procedures were performed. Pain levels were recorded at 4, 6, 8, 12, and 24 hours using the VAS scale to compare the effectiveness of postoperative ibuprofen with preoperative dexamethasone.
  Interventions: Drug: Ibuprofen group

INTERVENTIONS:
Drug: Dexamethasone 4 mg — Participants in this group received a single 4 mg oral dose of dexamethasone 1 hour before undergoing endodontic treatment. No additional preoperative analgesics were administered. Standard endodontic procedures, including local anesthesia, were performed. Post-treatment, no routine analgesic medication was provided unless additional pain relief was required. Pain intensity was assessed at 4, 6, 8, 12, and 24 hours using the Visual Analog Scale (VAS) to evaluate the efficacy of preoperative dexamethasone in controlling postoperative pain and inflammation.
  Arms: Dexamethasone Group
Drug: Ibuprofen group — Participants in this group received no preoperative medication but were prescribed 400 mg of ibuprofen every 4 hours postoperatively for pain management. The same standard endodontic procedures were performed. Pain levels were recorded at 4, 6, 8, 12, and 24 hours using the VAS scale to compare the effectiveness of postoperative ibuprofen with preoperative dexamethasone.
  Arms: Ibuprofen Group

SUMMARY:
This Phase IV randomized clinical trial (RCT) evaluated the efficacy of preoperative administration of a single 4 mg oral dose of dexamethasone in reducing postoperative pain and inflammation following endodontic treatment. Conducted at the Department of Endodontics, PhD Program, Faculty of Dentistry, University of Salamanca, the study included 82 participants who were randomly assigned to either the test group (preoperative dexamethasone) or the control group (postoperative ibuprofen 400 mg every 4 hours).

Pain intensity was measured using the Visual Analog Scale (VAS) at 4, 6, 8, 12, and 24 hours postoperatively. Results indicated significantly lower pain perception in the dexamethasone group compared to the ibuprofen group at all time points, with the majority of dexamethasone-treated patients reporting only mild pain. No adverse effects were observed in either group, and no patient required additional rescue analgesia.

The findings suggest that a single preoperative dose of dexamethasone is a safe and effective strategy for managing postoperative pain in endodontic procedures, providing superior analgesia compared to the standard postoperative ibuprofen regimen.

Keywords: Endodontic pain, dexamethasone, preoperative analgesia, randomized clinical trial, inflammation control, corticosteroids, endodontics.

DETAILED DESCRIPTION:
Background and Rationale:

Endodontic treatment is a standard dental procedure aimed at preserving teeth with irreversible pulp damage or infection. A common complication following such procedures is postoperative pain and inflammation, typically managed with nonsteroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen. However, corticosteroids like dexamethasone, known for their potent anti-inflammatory and analgesic properties, may offer an alternative approach.

Dexamethasone is a long-acting glucocorticoid that inhibits phospholipase A2, thereby reducing the production of prostaglandins and leukotrienes-key mediators in the inflammatory cascade. This mechanism potentially prevents peripheral sensitization and hyperalgesia, which are central to post-endodontic pain. While dexamethasone has shown efficacy in oral surgery, its use as a preoperative analgesic in endodontics remains under-investigated.

Study Objectives:

The primary objective is to evaluate whether a single 4 mg oral dose of dexamethasone administered preoperatively reduces postoperative pain following endodontic treatment. Secondary objectives include assessing the need for rescue analgesia and monitoring for adverse effects.

Study Design:

This is a Phase IV randomized clinical trial using a parallel assignment model with a 1:1 allocation ratio. The study was conducted at the Faculty of Dentistry, University of Salamanca.

Participants and Randomization:

A total of 82 adult patients (aged 20-50) requiring endodontic intervention were enrolled. Participants were randomized into two groups:

Dexamethasone Group (Experimental): Received 4 mg dexamethasone orally 1 hour prior to the procedure.

Ibuprofen Group (Active Comparator): Received no preoperative medication but were prescribed 400 mg ibuprofen every 4 hours postoperatively.

Blinding:

The study was single-blind; participants were unaware of their group allocation.

Intervention:

All patients underwent standardized endodontic treatment involving local anesthesia, rubber dam isolation, mechanical root canal instrumentation using rotary systems, and irrigation with sodium hypochlorite. Root canal obturation followed standard protocols using gutta-percha and resin-based sealers.

Outcome Assessment:

Pain intensity will be measured using the Visual Analog Scale (VAS) at 4, 6, 8, 12, and 24 hours postoperatively. Secondary outcomes include the number of participants requiring rescue analgesia and any adverse effects reported during the first 24 hours.

Statistical Analysis:

Data will be analyzed using SPSS version 22.0. The normality of continuous variables will be assessed using the Shapiro-Wilk test. Pain intensity scores will be compared using ANOVA with Tukey post-hoc tests for multiple comparisons. A p-value < 0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be eligible for the study:
* Age Range: 20 to 50 years old.
* Indication for Endodontic Treatment: Patients requiring root canal therapy due to irreversible pulpitis (with or without apical lesion), pulp necrosis, retreatment with periapical lesion, or endodontic surgery.
* Eligible Teeth: Any dental group (anterior, premolar, molar, both maxillary and mandibular).
* General Health Status: Classified as ASA I (healthy individuals without systemic conditions) according to the American Society of Anesthesiologists (ASA) Physical Status Classification.
* Consent: Willingness to participate in the study and ability to provide signed informed consent.

Exclusion Criteria:

* Participants will be excluded if any of the following conditions apply:
* Age: Under 20 or over 50 years old.
* Medical Conditions:

Immunocompromised individuals (e.g., HIV/AIDS, cancer patients undergoing chemotherapy).

Systemic diseases such as diabetes mellitus, osteoporosis, acute psychosis, glaucoma, cataracts.

Patients with tuberculosis or systemic fungal infections. Gastrointestinal conditions such as ulcerative colitis, peptic ulcers, or diverticulitis.

-Medication Use: Use of NSAIDs or corticosteroids within 48 hours prior to the intervention. Regular use of barbiturates.

-Dental Factors: Tooth fractures involving the roots. Severe dental hypersensitivity that may interfere with pain assessment.

-Pregnancy and Lactation: Pregnant or breastfeeding women will be excluded due to potential effects of dexamethasone.

-Non-Compliance: Patients who decline participation or are unwilling to follow study procedures, including pain assessment and follow-up.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (Visual Analog Scale Score) | 4, 6, 8, 12, and 24 hours post-endodontic treatment
  Description: Pain intensity will be measured using the Visual Analog Scale (VAS), a 10-centimeter horizontal line where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Participants will mark their perceived pain levels at each time point to assess postoperative discomfort following endodontic treatment.
  Scale Range: 0 (no pain) to 10 (worst pain)
  Interpretation: Higher scores indicate a worse outcome (greater pain intensity).

SECONDARY OUTCOMES:
Need for Rescue Analgesia | 24 hours post-endodontic treatment
  Description: The number of participants requiring additional pain medication (rescue analgesia) beyond the assigned intervention will be recorded. This measure will help evaluate whether preoperative dexamethasone can reduce the necessity for additional analgesics compared to standard ibuprofen therapy.

OTHER OUTCOMES:
Adverse Effects | Up to 24 hours post-treatment
  Participants will be monitored for any adverse effects associated with dexamethasone or ibuprofen, including gastrointestinal discomfort, dizziness, nausea, allergic reactions, or other reported symptoms.
Gender-Based Pain Response | 4, 6, 8, 12, and 24 hours post-treatment
  Pain intensity VAS(Visual Analog Scale score) will be analyzed separately for male and female participants to determine whether there are gender-based differences in pain perception and response to dexamethasone and ibuprofen.
Inflammatory Symptoms | 24 hours post-treatment
  Participants will be asked to report swelling, redness, or localized discomfort at the treatment site to assess the anti-inflammatory effects of dexamethasone compared to ibuprofen.
Patient Satisfaction with Pain Management | 24 hours post-treatment
  Patients will rate their overall satisfaction with pain management on a Likert scale (1-5), with 1 being "very dissatisfied" and 5 being "very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Javier Flores- Fraile Supervisor PI, PhD in Surgery and Dentistry, Study Director — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No
The study does not plan to share individual participant data (IPD) due to patient confidentiality and ethical considerations. Only aggregated, anonymized data will be presented in publications and reports.